CLINICAL TRIAL: NCT05630144
Title: Deprescribing for Older Adults After Hospital Discharge in Home Health Care - A Pilot Feasibility Study of the HomeMed Deprescribing Intervention
Brief Title: Deprescribing for Older Adults After Hospital Discharge in Home Health Care
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Rochester (Other)
Collaborators: National Institute on Aging (NIA) (NIH)
Responsible Party: Principal Investigator, Thomas Caprio, Professor - Department of Medicine, Geriatrics/Aging (SMD), University of Rochester
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: STUDY00007846; R24AG064025 (NIH)
Record Dates: First submitted 2022-11-17; First posted 2022-11-29 (Actual); Last update posted 2025-07-16 (Actual); Status verified 2025-07

CONDITIONS: Polypharmacy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- All Participants (Experimental)
  Interventions: Behavioral: HomeMed

INTERVENTIONS:
Behavioral: HomeMed — The HomeMed intervention is a multidisciplinary deprescribing intervention including home visits and team-based telehealth communication (optional). The components included in the HomeMed intervention include home medication review, medication education and provision of tools to assist the patients with medication administration, assessment of deprescribing targets by a trained geriatric clinical pharmacist, communication with the patient's treating primary care provider about deprescribing recommendation, deprescribing implementation (optional), and deprescribing monitoring (optional). Depending on the patient's treating primary care provider's decision on deprescribing and monitoring, the number of home visits ranges from a minimum of three to more with the entire duration of the intervention ranging from approximately 1 to 3 months.

SUMMARY:
The purpose of this study is to examine the feasibility of providing a medication optimization program to improve patient health outcomes during the transition from hospital to home. This is because the period after hospital discharge is critical to long-term recovery, overall quality of life, and prevention of future hospitalizations.

ELIGIBILITY:
Patient Inclusion Criteria:

* 65 years of age and older
* currently hospitalized or having been hospitalized in the previous 2 weeks
* having a discharge disposition of home with a referral to receive HHC services from URMHC, or currently receiving HHC services from URMHC
* taking more than 10 regular medications daily
* having a primary care provider who is in the URMC system
* Ability to self-consent
* English-speaking

Patient Exclusion Criteria:

* end-of-life prognosis in the following 6 months
* currently receiving hospice care, end-of-life care, or palliative care
* conditions that impact the receipt of the intervention, such as severe cognitive impairment that interferes with the subject's ability to communicate with interventionists;
* substantial difficulties in hearing, vision, and verbal expression that disable the participant from communicating effectively while receiving the HomeMed intervention

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 5 (Actual)
Dates: Start 2023-03-29 (Actual); Primary Completion 2025-05-30 (Actual); Study Completion 2025-05-30 (Actual)

PRIMARY OUTCOMES:
mean time spent on intervention | 3 months
number of participants who complete a post intervention survey about feasibility | 3 months
Percentage of participants undergoing deprescribing | 3 months
Percentage of intervention adherence indicators checked | 3 months
Percentage of patients who improve in ability to do things that are important before and after intervention | 3 months
Total number of medications used per participant | 3 months
Percentage of patients who report a reduction in medication burden | 3 months
  Medication burden will be reported by phone or survey.
Percentage of participants who report a reduction in medication side effect | 3 months
  Side effects will be collected by phone.

CONTACTS AND LOCATIONS:
Locations (1):
- University of Rochester Medical Center, Rochester, New York, United States

IPD SHARING:
Plan to Share IPD: No